CLINICAL TRIAL: NCT00000751
Title: A Phase III Randomized, Double-Blind, Controlled Study of the Use of Anti-HIV Immune Serum Globulin (HIVIG) for the Prevention of Maternal-Fetal HIV Transmission in Pregnant Women and Newborns Receiving Zidovudine (AZT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 185
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2006-05

CONDITIONS: HIV Infections; Pregnancy
Keywords: Pregnancy; Pregnancy Complications, Infectious; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine; Immunoglobulins, Intravenous; Immunization, Passive
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Immunoglobulins; Zidovudine

INTERVENTIONS:
Drug: Anti-HIV Immune Serum Globulin (Human)
Drug: Globulin, Immune
Drug: Zidovudine

SUMMARY:
To evaluate the effect of anti-HIV immune serum globulin (HIVIG) versus immune globulin (IVIG) administered during pregnancy and to the newborn, in combination with zidovudine (AZT) administered intrapartum and to the newborn, on incidence of HIV infection in infants born to HIV-infected women who received AZT during pregnancy for medical indications.

Vertical transmission of HIV from mother to child may occur before, during, or after parturition (via breast-feeding). It is believed that therapy administered both during pregnancy and intrapartum may help prevent vertical transmission. Additionally, adjunctive short-term antiretroviral therapy for the newborn, following the intensive viral exposure presumed to occur at birth, may be necessary.

DETAILED DESCRIPTION:
Vertical transmission of HIV from mother to child may occur before, during, or after parturition (via breast-feeding). It is believed that therapy administered both during pregnancy and intrapartum may help prevent vertical transmission. Additionally, adjunctive short-term antiretroviral therapy for the newborn, following the intensive viral exposure presumed to occur at birth, may be necessary.

Pregnant women who are currently receiving AZT are randomized at 20-30 weeks of gestation to begin receiving either HIVIG or IVIG every 28 days up to delivery. Within 12 hours after birth, the infant receives an infusion of matching study drug. During labor, all women receive an intravenous loading dose of AZT administered over 1 hour, followed by continuous infusion during the intrapartum period until the umbilical cord is clamped. All infants receive AZT syrup every 6 hours, beginning as soon as oral fluids are tolerated but within 8-12 hours after birth and continuing for 6 weeks. Women are followed until 26 weeks postpartum. Infants are followed at weeks 1, 2, 4, and then every 4 weeks through week 24, every 12 weeks through week 60, at week 78 (18 months), and at week 104 (24 months).

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Women - Medications as required for obstetrical management of HIV infection (e.g., acyclovir, ketoconazole, isoniazid, antibiotics, or other antiretroviral therapy if intolerant or failing on AZT), unless specifically excluded.
* Infants - Drug treatment for signs of drug withdrawal (phenobarbital, chlorpromazine, tincture of opium, paregoric or Valium).
* Infants - Medications as indicated for management of an HIV-exposed infant (e.g., hepatitis B vaccine, syphilis treatment, Pneumocystis carinii pneumonia prophylaxis).

Patients must have:

* Documented HIV infection.
* Been receiving AZT during current pregnancy for medical indications.
* Gestational age between 20 and 30 weeks.
* Intention to carry pregnancy to term.
* Available venous access (placement of central line or Hickman catheter not indicated for study purposes).
* Willingness to be followed by a participating site for study duration.

NOTE:

* Father of fetus (if available after a reasonable attempt to contact him) must also provide informed consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Illness associated with excessive protein loss, e.g., severe proteinuria (protein >= 4 g protein in a 24-hour urine collection).

Patients with the following prior conditions are excluded:

* Evidence of pre-existing fetal anomalies (e.g., anencephaly, renal agenesis, or Potter's syndrome) that may result in a high probability that the fetus-infant would not survive to the end of the study period.
* Chorionic villus sampling (CVS) or percutaneous umbilical blood sampling (PUBS) occurring in this pregnancy prior to study entry.
* Illness associated with excessive protein loss, e.g., chronic diarrhea with no documented weight gain in a 3-month period during pregnancy.
* Pre-existing conditions such as hypogammaglobulinemia or immune thrombocytopenia that are felt to require IVIG therapy.

Prior Medication:

Excluded:

* Receipt of anti-HIV vaccines or passive immunotherapy with HIVIG or IVIG during this pregnancy prior to study entry.
* Receipt of antiretroviral agents other than AZT during this pregnancy prior to study entry (e.g., rCD4, CD4-IgG, d4T, ddC, ddI).

Ages: 13 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1600
Dates: Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ER Stiehm, Study Chair; J Lambert, Study Chair
Locations (51):
- United States (48):
  - UCSD Med Ctr / Pediatrics / Clinical Sciences, La Jolla, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA Med Ctr / Pediatric, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - San Francisco Gen Hosp, San Francisco, California
  - UCSF / Moffitt Hosp - Pediatric, San Francisco, California
  - Denver Gen Hosp, Denver, Colorado
  - Children's Hosp of Denver, Denver, Colorado
  - Univ of Connecticut / Farmington, Farmington, Connecticut
  - Children's Hosp of Washington DC, Washington D.C., District of Columbia
  - Washington Hosp Ctr, Washington D.C., District of Columbia
  - Howard Univ Hosp, Washington D.C., District of Columbia
  - Univ of Florida Health Science Ctr / Pediatrics, Jacksonville, Florida
  - Univ of Miami (Pediatric), Miami, Florida
  - Univ of Illinois College of Medicine / Pediatrics, Chicago, Illinois
  - Tulane Univ / Charity Hosp of New Orleans, New Orleans, Louisiana
  - Univ Hosp, New Orleans, Louisiana
  - Univ of Maryland at Baltimore / Univ Med Ctr, Baltimore, Maryland
  - Johns Hopkins Hosp - Pediatric, Baltimore, Maryland
  - Children's Hosp of Boston, Boston, Massachusetts
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Boston City Hosp / Pediatrics, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Univ of Massachusetts Med School, Worcester, Massachusetts
  - Children's Hosp of Michigan, Detroit, Michigan
  - Univ of Medicine & Dentistry of New Jersey / Univ Hosp, Newark, New Jersey
  - Children's Hosp at Albany Med Ctr, Albany, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mount Sinai Med Ctr / Pediatrics, New York, New York
  - Columbia Presbyterian Med Ctr, New York, New York
  - State Univ of New York at Stony Brook, Stony Brook, New York
  - SUNY Health Sciences Ctr at Syracuse / Pediatrics, Syracuse, New York
  - Bronx Lebanon Hosp Ctr, The Bronx, New York
  - Univ of North Carolina at Chapel Hill / Duke Univ Med Ctr, Durham, North Carolina
  - Case Western Reserve Univ - Pediatric, Cleveland, Ohio
  - Children's Hosp of Philadelphia, Philadelphia, Pennsylvania
  - Hosp of the Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Saint Christopher's Hosp for Children, Philadelphia, Pennsylvania
  - Temple Univ School of Medicine, Philadelphia, Pennsylvania
  - Med Univ of South Carolina, Charleston, South Carolina
  - Regional Med Ctr at Memphis, Memphis, Tennessee
  - Methodist Hosp Central, Memphis, Tennessee
  - Saint Jude Children's Research Hosp of Memphis, Memphis, Tennessee
  - Children's Med Ctr of Dallas, Dallas, Texas
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Texas Children's Hosp / Baylor Univ, Houston, Texas
  - Children's Hospital & Medical Center / Seattle ACTU, Seattle, Washington
- Puerto Rico (3):
  - Ramon Ruiz Arnau Univ Hosp / Pediatrics, Bayamón
  - Univ of Puerto Rico / Univ Children's Hosp AIDS, San Juan
  - San Juan City Hosp, San Juan

REFERENCES:
- [Background] Mofenson LM. Interventions to reduce perinatal transmission. Natl Conf Women HIV. 1997 May 4-7:125 (abstract no 2011)
- [Background] McKinney RE Jr. Ongoing and future trials of antiretroviral therapy in the pediatric AIDS clinical trials group (PACTG). Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:173
- [Background] Lambert J, Fletcher C, Mofenson L, Stiehm ER, Moye J, Meyer W, Nemo G, Mathieson B, Hirsch G. Pharmacokinetics (PK) of hyperimmune HIV immunoglobulin (HIVIG) in HIV+ pregnant females & newborns. Natl Conf Hum Retroviruses Relat Infect (2nd). 1995 Jan 29-Feb 2:148
- [Background] Lambert JS, Watts DH, Mofenson L, Stiehm ER, Harris DR, Bethel J, Whitehouse J, Jimenez E, Gandia J, Scott G, O'Sullivan MJ, Kovacs A, Stek A, Shearer WT, Hammill H, van Dyke R, Maupin R, Silio M, Fowler MG. Risk factors for preterm birth, low birth weight, and intrauterine growth retardation in infants born to HIV-infected pregnant women receiving zidovudine. Pediatric AIDS Clinical Trials Group 185 Team. AIDS. 2000 Jul 7;14(10):1389-99. doi: 10.1097/00002030-200007070-00012. PMID 10930154
- [Background] Mofenson LM, Lambert JS, Stiehm ER, Bethel J, Meyer WA 3rd, Whitehouse J, Moye J Jr, Reichelderfer P, Harris DR, Fowler MG, Mathieson BJ, Nemo GJ. Risk factors for perinatal transmission of human immunodeficiency virus type 1 in women treated with zidovudine. Pediatric AIDS Clinical Trials Group Study 185 Team. N Engl J Med. 1999 Aug 5;341(6):385-93. doi: 10.1056/NEJM199908053410601. PMID 10432323
- [Background] Lambert JS, Mofenson LM, Fletcher CV, Moye J Jr, Stiehm ER, Meyer WA 3rd, Nemo GJ, Mathieson BJ, Hirsch G, Sapan CV, Cummins LM, Jimenez E, O'Neill E, Kovacs A, Stek A. Safety and pharmacokinetics of hyperimmune anti-human immunodeficiency virus (HIV) immunoglobulin administered to HIV-infected pregnant women and their newborns. Pediatric AIDS Clinical Trials Group Protocol 185 Pharmacokinetic Study Group. J Infect Dis. 1997 Feb;175(2):283-91. doi: 10.1093/infdis/175.2.283. PMID 9203648
- [Background] Lambert JS, Moye J, Sapan C, Mofenson L, Fletcher C, Whitehouse J, Fowler MG, Nemo G, Stiehm ER. Demonstration of feasibility and preliminary safety and pharmaco-kinetics in a phase III study of hyperimmune HIV intravenous immunoglobulin (HIV-IG) to prevent maternal-fetal HIV transmission. Int Conf AIDS. 1996 Jul 7-12;11(2):84 (abstract no WeB3163)
- [Background] Frenkel LM. Therapeutic issues pertaining to HIV-1 infected pregnant women in developed countries. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sept 26-29
- [Background] Watts DH, Lambert J, Stiehm ER, Harris DR, Bethel J, Mofenson L, Meyer WA 3rd, Mathieson B, Fowler MG, Nemo G; PACTG 185 Study Team. Progression of HIV disease among women following delivery. J Acquir Immune Defic Syndr. 2003 Aug 15;33(5):585-93. doi: 10.1097/00126334-200308150-00006. PMID 12902802
- [Result] Lambert JS. HIV vaccines in infants and children. Paediatr Drugs. 2005;7(5):267-76. doi: 10.2165/00148581-200507050-00001. PMID 16220994